CLINICAL TRIAL: NCT02298244
Title: Safety Procedure Pulmonary Artery Denervation in Addition to Pulmonary Vein Isolation Combined With Ganglionated Plexi Ablation in Patients With Persistent Atrial Fibrillation and Pulmonary Hypertension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Krasnoyarsk Regional Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PDPVI16112014
Record Dates: First submitted 2014-11-16; First posted 2014-11-21 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-11

CONDITIONS: Atrial Fibrillation; Hypertension, Pulmonary; Heart Diseases; Arrhythmias, Cardiac; Pathologic Processes; Cardiovascular Diseases; Lung Diseases
Keywords: Pulmonary Hypertension; Atrial Fibrillation; Pulmonary Arterial Denervation; Safety; Pulmonary Arterial GP Ablation
MeSH Terms: conditions — Atrial Fibrillation; Hypertension, Pulmonary; Heart Diseases; Arrhythmias, Cardiac; Pathologic Processes; Cardiovascular Diseases; Lung Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- PV isolation + GP Ablation (Active Comparator)
  Interventions: Procedure: PV isolation + GP Ablation
- PV isolation + GP ablation + Pulmonary GP ablation (Active Comparator)
  Interventions: Procedure: PV isolation + GP ablation + Pulmonary GP ablation

INTERVENTIONS:
Procedure: PV isolation + GP Ablation — In real time builds the 3D card LA using nonfluoroscopic navigation system.Left and right PVs encircle in 1 lesion line by circumferential PV isolation.Radiofrequency energy delivered at 43◦C,35 W,0.5 cm away from the PV ostia at the anterior wall,and reduced to 43◦C,30 W,1 cm away from the PV ostia at the posterior wall,with a saline irrigation speed of 17 ml/min.Each lesion of ablation continuously until the local potential amplitude decreased by >80% or RF energy deliveries exceeded 40 seconds.The endpoint of circumferential PV isolation is PV isolation;this confirm when Lasso mapping show the disappearance of all PV potentials or the dissociation of PV potentials from left atrial activity.To accomplish ganglionated plexi ablation,LA target sites were identified as the anatomic locations where vagal reflexes were evoked by transcatheter HFS.Rectangular electrical stimuli were delivered at a frequency of 50 Hz,output amplitude 15V and pulse duration of 10 ms,for 5 sec
  Arms: PV isolation + GP Ablation
Procedure: PV isolation + GP ablation + Pulmonary GP ablation — The procedure of AF ablation is the same like in the circumferential PV isolation + GP Ablation.
  8-Fr sheath is carried through the right heart into the pulmonary artery trunk. Using ablation electrode constructed 3D map of the pulmonary artery trunk and the right and left main branches. Further HFS performed with the tip ablation electrode at the bifurcation of the pulmonary artery and in the ostium of the left and right pulmonary arteries (less than 2 mm distal to the bifurcation) 20 Hz, duration of each stimulus 10 ms. A positive response would be considered an increase in the RR interval of more than 50% of baseline within 10 seconds. In areas with a positive response to HFS, will be performed RFA Efficiency criterion: no previously described responses to HFS in the ablation area. Parameters RFA: 8-10 watts for 60 seconds duration at one point, the irrigation speed of 5 ml / min.
  Arms: PV isolation + GP ablation + Pulmonary GP ablation

SUMMARY:
Some patients with a long history of AF develops PH "reactive" type with an increase in pulmonary vascular resistance due to vasoconstriction or structural changes of the vascular wall. RFA PVI + RFA GP is the "gold standard" in the treatment of patients with persistent AF, do not respond to optimal therapy. The rear area of the pulmonary artery bifurcation is adjacent to the roof and part of the front of the left atrium. In the projection of this area are ganglionic plexus of the left atrium, the sympathetic nerve fibers of the pulmonary artery and baroreceptors main pulmonary artery.Recent studies have shown that radiofrequency denervation of the pulmonary artery improves the quality of life in patients with PH.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic, drug - refractory AF ( inefficiency 1C or III Class antiarrhythmic drugs), history of AF 6 months or more without the restoration of sinus rhythm.
* MPAP ≥25 mmHg
* PCWP≥15 mmHg
* Pulmonary vascular resistance (PVR). The PVR =(mPAP-PCWP)/ carbon monoxide] > 2.5 woods unit

Exclusion Criteria:

* Left ventricular ejection fraction <35%
* Diameter LA> 60 mm on transthoracic echocardiography in the "M" -Mode or volume of LA more than 140 ml
* Significant regurgitation at the mitral valve
* Uncorrected congenital heart disease
* RFA PVI, RFA GP, PADN in history
* Foregoing heart surgery
* Life expectancy less than 12 months
* WHO group I, III, IV, V pulmonary artery hypertension
* Tricuspid valve stenosis, pulmonary supravalve stenosis.
* Cancer
* Pregnancy
* Thromboembolism LA history
* Hyperthyroidism.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
death | 6 months
  all-cause death at 1, 3, 6 months after procedure
Perioperative Complications | 6 months
  perforation / dissection at any level, an acute thrombosis in the pulmonary artery, re - hospitalization due to Pulmonary Hypertension, Atrial Fibrillation) immediately after and at 1, 3, 6 months after procedure

SECONDARY OUTCOMES:
Mean Pulmonary Artery Pressure | 6 months
  Measured by cardiac echo at 1,3,6 months
recurrence of AF / AFL / AT | 6 months
  Measured by 48-hours ECG at 1,3,6 months
Quality of life | 6 months
  Measured by SF-36 at 1, 6 months
6-minute walk distance | 6 months
  Measured at 1,3,6 months
Pulmonary vascular resistance | 1 month
  Measured by right heart catheterization; The PVR =(mPAP-PCWP)/ carbon monoxide
Assessment of respiratory function | 6 months
  Respiratory function tests at 1, 6 months